CLINICAL TRIAL: NCT02739308
Title: Effects of Proprioceptive Training on Neurofunctional Control and Ankle Sprains Incidence in Fencers: a Randomized Controlled Trial
Brief Title: Effects of Proprioceptive Training on Neurofunctional Control and Ankle Sprains Incidence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Gabriela Souza de Vasconcelos, Physical Therapy and Student of Post Graduate of UFRGS, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 436620
Record Dates: First submitted 2016-04-06; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Ankle Injuries
Keywords: proprioception; ankle sprain; fencing
MeSH Terms: conditions — Ankle Injuries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention: Proprioceptive Training (Experimental): The intervention will be the implementation of a proprioceptive training program for the fencing athletes in the intervention group.
  In this study the training program will be developed for 12 weeks and will be applied during the heating of the athletes, three times a week and the duration of each session is 30 minutes. Each week will be chosen three of the 14 exercises adapted for fencing athletes, and preferably one of each category. The categories have exercises with different levels of difficulty and can change the exercises occur by different proposed levels or the complexity of the exercise by changing category. The training program will be implemented by the same evaluator over the 12 weeks.
  Interventions: Other: Proprioceptive Training
- Control (Placebo Comparator): The control group will not make the intervention and will continue with the usual training fencing.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Proprioceptive Training — In this study the training program will be developed for 12 weeks and will be applied during the heating of the athletes , three times a week and the duration of each session is 30 minutes. Each week will be chosen three of the 14 exercises adapted for fencing athletes , and preferably one of each category.
  Arms: Intervention: Proprioceptive Training
Other: Control Group — The control group will not make the intervention and will continue with usual training fencing.
  Arms: Control

SUMMARY:
The aim of this study is to investigate the influence of a 12-week proprioceptive training program on the neurofunctional control and the incidence of ankle sprains in fencing athletes. The study will be developed in six stages: familiarization, pre intervention, intervention, post intervention follow-up of three and six months. In the pre intervention stage will evaluate muscle strength inverters, everter, dorsal plantar flexors and ankle flexors through the isokinetic dynamometer; the reaction time of these muscles during Lunge Test; neuromuscular control during the Star Excursion Balance Test and performance in Drop Vertical Jump Test. In the intervention athletes will perform proprioceptive training for 12 weeks, three times a week, lasting 30 minutes. In the post intervention, the follow up of three to six months will be held the same pre intervention of the tests and recording the incidence of injuries occurred during the study. The expected result at the end of the study is to improve all variables, increasing the performance of athletes and decreasing the incidence of ankle sprains.

DETAILED DESCRIPTION:
Fencing is an agility sport, with higher incidence of injuries in the lower limbs, with the ankle sprain the most prevalent. Injury prevention is very important to improve performance and reduce time off of athletes. Proprioceptive training programs can be added to the training of athletes, since in addition to the easy application and low cost, proprioception serves to stabilize the joint, preventing injuries. Therefore the aim of this study is to investigate the influence of a 12-week proprioceptive training program on the neurofunctional control and the incidence of ankle sprains in fencing athletes. The study will be a randomized clinical trial, with fencing athletes from 14 to 25, a multi-sport club of Porto Alegre/RS, and developed in six stages: familiarization, pre intervention, intervention, post intervention follow-up of three and six months. The first step will be to familiarize themselves with the force of testing and registration of injuries in the previous year. In the pre intervention stage will evaluate muscle strength inverters, everter, dorsal plantar flexors and ankle flexors through the isokinetic dynamometer; the reaction time of these muscles during Lunge Test; neuromuscular control during the Star Excursion Balance Test and performance in Drop Vertical Jump Test. In the intervention athletes will perform proprioceptive training for 12 weeks, three times a week, lasting 30 minutes. In the post intervention, the follow up of three to six months will be held the same pre intervention of the tests and recording the incidence of injuries occurred during the study. For statistical analysis, the data will be presented as mean and standard deviation and submitted to the Shapiro-Wilk test, ANOVA will be held for repeated measures and post hoc Bonferroni to determine differences. The effect size is calculated using Cohen's d test.o significance level is 0.05. The expected result at the end of the study is to improve all variables, increasing the performance of athletes and decreasing the incidence of ankle sprains.

ELIGIBILITY:
Inclusion Criteria:

* practicing fencing at least a year
* have between 14 and 30 years.

Exclusion Criteria:

* be in physical therapy or participating in prevention programs
* have damage to lower limbs that compromise the tests

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Onset muscle | 12 weeks
  The muscular reaction time will be assessed by electromyography during Lunge Test.

SECONDARY OUTCOMES:
Muscle Strength | 12 weeks
  The muscle strength of ankle will be assessed by isokinetic dynamometer.
Star Excursion Balance Test (SEBT) | 12 weeks
  The SEBT will be used to measure the dynamic neuromuscular control.
Drop Vertical Jump Test (DVJT) | 12 weeks
  The DVJT be used to assess the height of the heels, from surfaces 30, 40 and 50cm .
Cumberland Ankle Instability Tools (CAIT) | 12 weeks
  The CAIT will be used to assess whether the ankle has istabilidade
Injury questionnaire | 12 weeks
  This questionnaire will be used to assess the number of injuries and to joints they occurred.

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriela Souza de Vasconcelos, Porto Alegre, Rio Grande do Sul, Brazil